CLINICAL TRIAL: NCT01143636
Title: Investigation and Treatment of Central Nervous System Dysfunction in Chronic Pelvic Pain.
Brief Title: Transcranial Direct Stimulation in Chronic Pelvic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Felipe Fregni, Principal Investigator, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009-P-002048
Record Dates: First submitted 2010-04-20; First posted 2010-06-14 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Pain; Healthy
Keywords: Transcranial direct current stimulation; Chronic Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Transcranial Direct Current Stimulation; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: For the experiment in patients with pelvic pain, the design is parallel. For the experiment in healthy subjects, the design is crossover.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active tDCS - pelvic pain patients (Sham Comparator): ACTIVE tDCS: Subjects will receive a total of 10 consecutive sessions of active tDCS over a two-week period (administered Monday - Friday). During each session, the anode electrode will be placed over the primary motor cortex of the predominantly painful side.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS - pelvic pain patients (Experimental): SHAM tDCS: Subjects will receive a total of 10 consecutive sessions of sham tDCS over a two-week period (administered Mon-Fri). During each session, the anode will be placed over the primary motor cortex of the predominantly painful side.
  Interventions: Device: Transcranial Direct Current Stimulation
- Active tDCS - healthy (Experimental): The healthy controls will undergo one day of treatment with active tDCS. All participants will receive both active and sham stimulation in a randomized order.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham tDCS - healthy (Experimental): The healthy controls will undergo one day of treatment with sham tDCS. All participants will receive both active and sham stimulation in a randomized order.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Chronic pain subjects will be randomized to receive either active or sham stimulation for the duration of the trial. The subject will receive 10 consecutive sessions at an intensity of 2mA with each session lasting 20 minutes. If the subject receives active stimulation the current will be applied for the full 20 minutes, while in the sham group current will only be applied for 30 seconds. In the healthy cohort, subjects will receive one session of active stimulation and one session of sham stimulation. The parameters will be the same as the pain subjects, at an intensity of 2mA for 20 minutes.
  Other Names: tDCS, electrical stimulation

SUMMARY:
The purpose of this study is to determine whether transcranial direct current stimulation (tDCS) is effective in reducing pain in subjects with chronic pelvic pain. Our hypothesis is that tDCS will decrease pain significantly when compared to sham stimulation.

DETAILED DESCRIPTION:
The study encompasses two experiments: The first one involves patients with chronic pain, receiving 10 sessions of stimulation, active or sham (parallel design).

The second experiment involves involves healthy subjects, receiving active or sham tDCS over the primary motor cortex (crossover design).

ELIGIBILITY:
Inclusion Criteria:

1. Providing informed consent to participate in the study
2. 18 to 64 years old
3. Having symptoms of pelvic pain for more than 6 months with an average of 3 on a 0-10 VAS scale (for pelvic pain subjects only)
4. No history of or current genitourinary tuberculosis as self reported
5. No history of urethral cancer as self reported
6. No history or current bladder malignancy, high grade dysplasia or carcinoma in situ as self reported
7. No occurrence of ovarian, vaginal or cervical cancer in the previous 3 years as self reported
8. No current vaginal infection as self reported
9. No active herpes in previous 3 months as self reported
10. No antimicrobials for urinary tract infections in previous 3 months as self reported
11. Never treated with cyclophosphamide as self reported
12. No radiation cystitis as self reported
13. No neurogenic bladder dysfunction (due to a spinal cord injury, stroke, Parkinson's disease, multiple sclerosis, spina bifida or diabetic cystopathy) as self reported
14. Absence of bladder, ureteral or urethral calculi for previous 3 months as self reported
15. No urethritis for previous 3 months as self reported
16. No urethral dilatation, cystometrogram, bladder cystoscopy with full anesthesia or bladder biopsy in previous 3 months as self reported
17. Must not be pregnant
18. Eligible to MRI according to MRI screening checklist
19. No contraindications to tDCS:
20. No history of alcohol or drug abuse within the past 6 months as self reported
21. No use of carbamazepine as self reported
22. Does not have severe depression (with a score of >30 in the Beck Depression Inventory)
23. No history of neurological disorders as self reported
24. No history of unexplained fainting spells as self reported,
25. No history of head injury resulting in more than a momentary loss of consciousness as self reported
26. Have had no neurosurgery as self reported
27. No history of psychological disorders as self reported
28. Must have the ability to feel pain as self reported

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Fregni, MD, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pelvic Pain, Active tDCS: Experimental Group: Subjects received a total of 10 consecutive sessions of active tDCS over a two-week period (administered Monday - Friday). During each session, the anode electrode was placed over the primary motor cortex of the predominantly painful side. tDCS was delivered for 20 minutes at an intensity of 2mA. In the active group current was applied for the full 20 minutes.
- Pelvic Pain, Sham tDCS: Sham Comparator: Subjects received a total of 10 consecutive sessions of sham tDCS over a two-week period (administered Mon-Fri). During each session, the anode was placed over the primary motor cortex of the predominantly painful side. Each tDCS session lasts 20 minutes. However, during sham stimulation current was only applied for 30 seconds at an intensity of 2mA.
- Healthy Controls: Active tDCS/Sham tDCS: Healthy Controls: These subjects received one single session of active tDCS and one one single session of sham tDCS. There was a time interval of at least one week in between the randomized stimulation sessions to prevent a carryover effect. This group received active stimulation first. Subjects received stimulation for 20 minutes at an intensity of 2mA. In the sham condition, current was only applied for the first 30 seconds and remained off for the rest of the 20 minute period.
- Healthy Subjects: Sham tDCS/Active tDCS: Healthy Controls: These subjects received one single session of sham tDCS and one single session of active tDCS. There was a time interval of at least one week in between the randomized stimulation sessions to prevent a carryover effect. This group received sham stimulation first. Subjects received stimulation for 20 minutes at an intensity of 2mA. In the sham condition, current was only applied for the first 30 seconds and remained off for the rest of the 20 minute period.
Period: Overall Study
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS | Healthy Controls: Active tDCS/Sham tDCS | Healthy Subjects: Sham tDCS/Active tDCS
Started | 6 | 5 | 8 | 7
Completed | 5 | 4 | 8 | 7
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active tDCS - Pelvic Pain: Experimental Group: Subjects received a total of 10 consecutive sessions of active tDCS over a two-week period (administered Monday - Friday). During each session, the anode electrode was placed over the primary motor cortex of the predominantly painful side. tDCS was delivered for 20 minutes at an intensity of 2mA. In the active group current was applied for the full 20 minutes.
- Sham tDCS - Pelvic Pain: Sham Comparator: Subjects received a total of 10 consecutive sessions of sham tDCS over a two-week period (administered Mon-Fri). During each session, the anode was placed over the primary motor cortex of the predominantly painful side. Each tDCS session lasts 20 minutes. However, during sham stimulation current was only applied for 30 seconds at an intensity of 2mA.
- Active tDCS&Sham tDCS - Healthy Controls: Healthy Controls: These subjects received one single session of active tDCS and one one single session of sham tDCS. There was a time interval of at least one week in between the randomized stimulation sessions to prevent a carryover effect. This group received active stimulation first. Subjects received stimulation for 20 minutes at an intensity of 2mA. In the sham condition, current was only applied for the first 30 seconds and remained off for the rest of the 20 minute period.
- Total: Total of all reporting groups
Arm/Group | Active tDCS - Pelvic Pain | Sham tDCS - Pelvic Pain | Active tDCS&Sham tDCS - Healthy Controls | Total
Number analyzed (Participants) | 6 | 5 | 15 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 5 | 15 | 26
  >=65 years | 0 | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: participants]
  Female | 5 | 4 | 9 | 18
  Male | 1 | 1 | 6 | 8
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Pain Assessment
Description: We use the Visual analogue scale (VAS) to measure pain. The VAS is ranged from 0 to 10, with 0 reffering to no pain and 10 reffering the the worst possible pain. We used the difference between post treatment minus baseline to compare the two treatments (active versus sham tDCS).
Time Frame: baseline and at 2 weeks
Population: The VAS is performed in patients with pelvic pain (Experiment 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pelvic Pain, Active tDCS: Experimental Group: Subjects received a total of 20 consecutive sessions of active tDCS over a four-week period (administered Monday - Friday). During each session, the anode electrode was placed over the primary motor cortex of the predominantly painful side. tDCS was delivered for 20 minutes at an intensity of 2mA. In the active group current was applied for the full 20 minutes.
- Pelvic Pain, Sham tDCS: Sham Comparator: Subjects received a total of 20 consecutive sessions of sham tDCS over a four-week period (administered Mon-Fri). During each session, the anode was placed over the primary motor cortex of the predominantly painful side. Each tDCS session lasts 20 minutes. However, during sham stimulation current was only applied for 30 seconds at an intensity of 2mA.
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | -2.375 (1.79) | -1.625 (2.46)

2. Primary Outcome: Pressure Pain Threshold
Description: Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain.
  The change in pressure pain threshold (post minus pre intervention) is use for the analysis.
Time Frame: baseline and at 2 weeks
Population: The pain pressure test is performed in healthy participants (exp 2).
Measure: Mean (Standard Deviation); unit: lb
Groups:
- Healthy Controls: Active tDCS: Healthy Controls: These subjects received one single session of active tDCS and one one single session of sham tDCS. There was a time interval of at least one week in between the randomized stimulation sessions to prevent a carryover effect. This group received active stimulation first. Subjects received stimulation for 20 minutes at an intensity of 2mA. In the sham condition, current was only applied for the first 30 seconds and remained off for the rest of the 20 minute period.
- Healthy Subjects: Sham tDCS: Healthy Controls: These subjects received one single session of sham tDCS and one single session of active tDCS. There was a time interval of at least one week in between the randomized stimulation sessions to prevent a carryover effect. This group received sham stimulation first. Subjects received stimulation for 20 minutes at an intensity of 2mA. In the sham condition, current was only applied for the first 30 seconds and remained off for the rest of the 20 minute period.
Arm/Group | Healthy Controls: Active tDCS | Healthy Subjects: Sham tDCS
Number analyzed (Participants) | 15 | 15
lb | 1.25 (0.75) | -1 (0.5)

3. Secondary Outcome: Quality of Life Scale (QOLS)
Description: The questionnaire on quality of life was performed at the end of the treatment session and compared between the two groups (active and sham) in patients with pelvic pain (Exp. 1). The QOLS has 16 items (total scores ranging from 16 to 112) the highest scores corresponding the best QOL.
Time Frame: 2 weeks
Population: We compared active and sham groups (Exp. 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 81.2 (15.4) | 78 (11.43)

4. Secondary Outcome: Clinical Global Impression - CGI
Description: This scale measures illness severity and was performed on patients with pelvic pain (Exp. 1). The scale was performed at end of the treatment and compared between the two groups (real and sham). The scale is divided in 3 sub-scales: Severity of illness (0-7), global improvement (0-7) and efficacy index (0-16), total scores ranging from 0 to 30. The highest scores corresponding to lowest clinical improvement.
Time Frame: 2 weeks
Population: Patients with pelvic pain (Exp 1)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 2.8 (0.4) | 3.3 (1.2)

5. Secondary Outcome: Visual Analogue Scale - Anxiety.This Scale Measures Patients' Level of Anxiety on a Scale (0-no Anxiety to 10-worst Anxiety Ever). It Was Performed at the End of the Treatment and Compared Between the 2 Groups (Real and Sham) in Patients With Pelvic Pain
Description: The scale was performed at the end of the treatment and compared between the 2 groups (real and sham) in patients with pelvic pain (Exp. 1).
Time Frame: 2 weeks
Population: This outcome measure was performed in patients with pelvic pain (Exp 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 0.8 (0.9) | 2.5 (2.1)

6. Secondary Outcome: Mini Mental Scale - MMS
Description: This scale measures patients cognitive impairment. It was performed at the end of the treatment and compared between the 2 groups (real and sham) in patients with pelvic pain (Exp. 1). It is a 30 points scale (total scores ranging from 0 to 30), the highest score corresponds to the highest cognitive status.
Time Frame: 2 weeks
Population: Patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 29.4 (0.8) | 28.75 (1.1)

7. Secondary Outcome: Beck Depression Inventory - BDI.
Description: BDI is a questionnaire used for detecting depression. It was performed at the end of the treatment and compared between the 2 groups (real and sham) in patients with pelvic pain (Exp. 1). It is a 21-question multiple-choice self-report inventory (scores ranging from 0 to 63 - 0 corresponds to no symptom of depression).
Time Frame: 2 weeks
Population: Patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 10 (9.7) | 6.75 (6.8)

8. Secondary Outcome: Patient Global Assessment - PGA
Description: This scale measures patient's assessment of general health. It was performed at the end of the treatment and compared between the 2 groups (real and sham) in patients with pelvic pain (Exp 1). The patient has to answer the question "how is your health overall" on a scale going from 0 to 10 (0 being the worst, 10 being the best).
Time Frame: 2 weeks
Population: Patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
units on a scale | 2.8 (0.9) | 2.75 (1.3)

9. Secondary Outcome: Von Frey
Description: This test is used to test subjects' sensitivity to a mechanical stimulus. It was performed before and and after the treatment and the difference (post minus pre) was compared between the 2 groups (real and sham) in patients with pelvic pain (Exp. 1). A set of filaments, typically from 0.008 grams force up to 300 grams force, is applied on the patients' skin. The mechanical threshold is defined as the moment when the patient detects the stimulus.
Time Frame: baseline and at 2 weeks
Population: Patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
grams | 0.7 (0.76) | -0.29 (0.48)

10. Secondary Outcome: Pain Pressure Threshold Test - PPT
Description: Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain.This test was applied before and after the treatment and the difference (post minus pre) was compared between the 2 groups (real and sham) in patients with pelvic pain (Exp 1).
Time Frame: baseline and at 2 weeks
Population: Patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
lb | 2.21 (3.93) | 1.41 (2.31)

11. Secondary Outcome: Diffuse Noxious Inhibitory Controls - DNIC.
Description: DNIC occurs when response from a painful stimulus (pain pressure threshold - PPT) is inhibited by another noxious stimulus (cold water). The difference between baseline and post treatment was compared between the 2 groups (real and sham) in patients with pelvic pain (Exp. 1).
Time Frame: baseline and at 2 weeks
Population: patients with pelvic pain (Exp. 1).
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Pelvic Pain, Active tDCS | Pelvic Pain, Sham tDCS
Number analyzed (Participants) | 5 | 4
lb | 2.46 (4.84) | 0.66 (2.39)

ADVERSE EVENTS:
Groups:
- SHAM tDCS - Pelvic Pain Patients: SHAM tDCS: Subjects will receive a total of 10 consecutive sessions of sham tDCS. During each session, the anode electrode will be placed on the primary motor cortex of the predominant painful side.
  For sham-controlled tDCS subjects, the current will be applied only for 30 seconds.
  Transcranial Direct Current Stimulation: Stimulation will be given at 2 mA for a period of 20 minutes.
- ACTIVE tDCS - Pelvic Pain Patients: ACTIVE tDCS: Subjects will receive a total of 10 consecutive sessions of active tDCS. During each session, the anode electrode will be placed on the primary motor cortex of the predominant painful side.
  Transcranial Direct Current Stimulation: Stimulation will be given at 2 mA for a period of 20 minutes.
- SHAM tDCS - Healthy: SHAM tDCS: Subjects will receive a single session of sham tDCS. The anode electrode will be placed on the primary motor cortex.
  For sham-controlled tDCS subjects, the current will be applied only for 30 seconds.
  Transcranial Direct Current Stimulation: Stimulation will be given at 2 mA for a period of 20 minutes.
- ACTIVE tDCS - Sham: ACTIVE tDCS: Subjects will receive a single session of active tDCS. The anode electrode will be placed on the primary motor cortex.
  Transcranial Direct Current Stimulation: Stimulation will be given at 2 mA for a period of 20 minutes.
Arm/Group | SHAM tDCS - Pelvic Pain Patients | ACTIVE tDCS - Pelvic Pain Patients | SHAM tDCS - Healthy | ACTIVE tDCS - Sham
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/4 | 5/5 | 11/15 | 15/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SHAM tDCS - Pelvic Pain Patients (N=4) | ACTIVE tDCS - Pelvic Pain Patients (N=5) | SHAM tDCS - Healthy (N=15) | ACTIVE tDCS - Sham (N=15)
Tingling (Skin and subcutaneous tissue disorders) | 3 | 5 | 10 | 11
Headache (Nervous system disorders) | 1 | 1 | 1 | 1
Neck pain (Nervous system disorders) | 1 | 1 | 0 | 0
Skin redness (Skin and subcutaneous tissue disorders) | 2 | 4 | 8 | 7
Sleepiness (Nervous system disorders) | 1 | 3 | 6 | 5
Diziness (Nervous system disorders) | 2 | 0 | 0 | 0
Scalp burning sensation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Trouble concentrating (Nervous system disorders) | 0 | 1 | 0 | 0
Acute mood change (Nervous system disorders) | 0 | 1 | 0 | 0
Nausea (General disorders) | 0 | 1 | 0 | 0
Itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No